CLINICAL TRIAL: NCT03855813
Title: Intra and Inter Reliability of 30 Seconds Chair Stand Test as Self-test for Patients With Knee Osteoarthritis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 255331_reliability30CST
Record Dates: First submitted 2019-02-24; First posted 2019-02-27 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2022-10

CONDITIONS: Osteoarthritis, Knee
Keywords: 30 seconds chair stand test; Performance test; Reliability
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Patients with knee osteoarthritis will perform the 30 seconds chair stand test as a self-test twice at home to evaluate intra rater reliability. Same patients will be tested with the same performance test by a physical therapist to evaluate the inter rater reliability.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test-retest reliability (Other): Patients with knee osteoarthritis will perform the 30 seconds chair stand test as a self test twice at home to evaluate intra rater reliability. Same patients will be tested with the same performance test by a physical therapist to evaluate the inter rater reliability.
  Interventions: Other: Intra rater reliability; Other: Inter rater reliability

INTERVENTIONS:
Other: Intra rater reliability — Patients will perform the 30 seconds chair stand test as a self-test twice at home with approximately two days apart. The last self-test should be performed approximately one week before the testing with a physical therapist.
Other: Inter rater reliability — Same patients performing the self-test will be tested by a physical therapist approximately one week after the last self-test. The physical therapist will be blind to the self-test results.

SUMMARY:
Background: It is estimated that 14% of the Swedish population have knee osteoarthritis. Common osteoarthritis symptoms are pain, stiffness and impaired physical function. To evaluate muscle strength in the lower extremities could indicate if there is a risk for a patient with osteoarthritis to worsen their disease. Increased muscle strength could improve physical function and pain for this patient group. A reliable self-test to evaluate physical function could help patients with diagnosed or suspected knee osteoarthritis to seek healthcare in time. The 30 seconds chair stand test (30 CST) is part of a test battery which is recommended to use for patients with osteoarthritis, both in research and in a clinical setting. It is a valid and a reliable measurement for patients with osteoarthritis. However, reliability studies of the 30 CST as a self-test is lacking.

Objective: To determine whether 30 CST is a reliable self-test to evaluate physical function among patients with knee osteoarthritis, we want to explore how much it differs in the test results when the patient is performing the test by herself and also compare it with when it is conducted in a clinical setting.

Methods: 147 participants with knee osteoarthritis will be recruited from three rehabilitations centers in primary care. The participant will perform the self-test twice at home, and the self-test will be compared with when the test is guided by a physical therapist at a rehabilitation center. The reliability results will be presented with an intraclass correlation coefficient and standard error measurement.

Estimated results: It is expected that the results from this study will clarify if 30 CST can be used as a self-test for persons with suspected or diagnosed/confirmed knee osteoarthritis. If this performance test show enough reliability to be used as a self-test, it could be used as an indicator if the patient should seek healthcare or not due to impaired function. To seek healthcare in an earlier phase usually require less efforts and often leads to shorter healthcare process. These improvements of the healthcare process could be of value to manage the expected future increase of osteoarthritis consultations to primary care.

DETAILED DESCRIPTION:
The project leader will be visiting recruiting units to inform and educate about the study protocol and data collection procedure.

Patient recruitment

Patients with knee osteoarthritis will be recruited from three rehabilitations centers in region Västra Götaland, Sweden. When eligible participants have been identified according to inclusion criteria, the participants will get written information about the study, including informed consent, manual to the 30 CST self-test, and questionnaires.

Data Collection

30 CST: The 30 CST will be performed on an approximately 45 cm high chair without armrest (if possible). The participant will be asked to perform as many stands as possible during 30 seconds. Start position is sitting on the chair, and the arms should be crossed over the chest during the whole test. The stands must be to upright standing position (i.e. fully extended hips and knees), and back to sitting position. The patients pain intensity will be measured with numeric rating scale before and during the test.

Manual to the 30 CST self-test and questionnaires: The participants will get a description of how the self-test should be performed. The self-test should be performed twice with approximately two days apart, and the last measurement should be approximately one week before the planned physical therapist testing with the 30 CST. The self-test results will be sealed in an envelope together with the completed questionnaires (demographic data, Intermittent and Constant Osteoarthritis Pain (ICOAP), Knee injury and Osteoarthritis Outcome Score (KOOS-PS)). The patients will be bringing these data to their physical therapists till their next visit at the rehabilitation center.

Physical therapist testing: All physical therapists in the study will get an education about the study protocol and the 30 CST. The physical therapists will be blind of the self-test result during the testing. They will use the same manual for the 30 CST as the patients. Participants will be notified how well their 30 CST test results are compared to the normal population. The participants' length and weight will be measured by the physical therapist to calculate the body mass index.

Reporting for adverse events

If the patients or physical therapists have to cancel the test, they will be able to report the reason why they needed to cancel (e.g. increased pain, unsafe due to difficulties with patients balance).

Data management

All data will be coded and managed according to the General Data Protection Regulation. All data will be confidential and only authorized will have access to the patient registry. No individual information can be identified since the results will be presented at group level. Data will be saved for at least 10 years to enable audit.

Sample size

Sample size was calculated with statistical software program PASS 16. A sample size of 117 participants with two observations per participant for inter respectively intra rater reliability achieved a power of 80% to detect an intraclass correlation coefficient (ICC) of 0.8 with a significance level of 0.05. With an estimated 20% drop-out rate, 147 participants are planned to be recruited to the study.

Statistical analysis

Demographic data will be analyzed descriptively. It will be presented as number and percent, mean and standard deviation, and median and 25th to 75th percentiles. Relative reliability (inter and intra reliability) will be presented with an ICC using a 95% confidence interval. ICC-values > 0.8 indicate enough reliability and values > 0.9 represent optimal reliability. Absolute reliability will be presented with standard error measurement. The analyses will be made in SPSS with a significance level of p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with knee osteoarthritis. The patients should have most problem with their knees, but are allowed to have osteoarthritis in other lower extremity joints.
* Independent in walking, with or without walking aids.
* Understand test instructions verbally and in writing.

Exclusion Criteria:

* Neurological disorders that affects the patients balance or gait.
* Severe somatic or mental illness that affect the physical functional performance or the ability to understand test instructions verbally or in text.
* Knee or hip replacement the past six months.
* Other knee surgery the past six months that could affect the physical functional performance.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2019-02-27 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-07-25 (Actual)

PRIMARY OUTCOMES:
30 seconds chair stand test as self-test. | Two occasions within approximately three days to establish intra rater reliability
  30 seconds chair stand test will be used as a self-test. Number of stands will be counted.
30 seconds chair stand test, comparison self-test vs clinical test. | Two occasions within approximately seven days to establish inter rater reliability
  30 seconds chair stand test will be used as a self-test and as a clinical test led by a physical therapist. Number of stands will be counted.

SECONDARY OUTCOMES:
Pain intensity during 30 seconds chair stand test | Three occasions within approximately 14 days, between the first and last testing with 30 seconds chair stand test.
  Pain intensity will be measured before and during the chair stand test with numeric rating scale between 0-10, where 0 means no pain and 10 worst imaginable pain.
Osteoarthritis pain | Baseline
  Osteoarthritis pain will be measured with Measure of Intermittent and Constant Osteoarthritis Pain: ICOAP. The questionnaire consists of two subscales, a) constant pain and b) intermittent pain. The total score ranges between 0 to 100 where 0 means no pain and 100 means extreme pain.
Difficulties with activities due to knee pain | Baseline
  Expericences of difficulties with activities due to patients knee pain will be measured with short version of Knee injury and Osteoarthritis Outcome Score (KOOS-PS). The total score ranges between 0-100 where 0 is great difficulties and 100 is no difficulties.

OTHER OUTCOMES:
Demographic data | Baseline
  Demographic data such as age, sex, body mass index (BMI), duration osteoarthritis diagnosis, other diseases, education level, origin, pain location, pain duration (knee). Patients' body weight and height will be measured to calculate the BMI.

CONTACTS AND LOCATIONS:
Overall Officials: Lena Nordeman, RPT, PhD, Principal Investigator — Research & Development Centre Södra Älvsborg
Locations (3):
- Sweden (3):
  - Närhälsan Lidköping Rehabmottagning, Lidköping, Västra Götaland County
  - Närhälsan Skara Rehabmottagning, Skara, Västra Götaland County
  - Närhälsan Trollhättan Rehabmottagning, Trollhättan, Västra Götaland County

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dobson F, Hinman RS, Roos EM, Abbott JH, Stratford P, Davis AM, Buchbinder R, Snyder-Mackler L, Henrotin Y, Thumboo J, Hansen P, Bennell KL. OARSI recommended performance-based tests to assess physical function in people diagnosed with hip or knee osteoarthritis. Osteoarthritis Cartilage. 2013 Aug;21(8):1042-52. doi: 10.1016/j.joca.2013.05.002. Epub 2013 May 13. PMID 23680877
- [Background] Jones CJ, Rikli RE, Beam WC. A 30-s chair-stand test as a measure of lower body strength in community-residing older adults. Res Q Exerc Sport. 1999 Jun;70(2):113-9. doi: 10.1080/02701367.1999.10608028. PMID 10380242
- [Background] Hawker GA, Davis AM, French MR, Cibere J, Jordan JM, March L, Suarez-Almazor M, Katz JN, Dieppe P. Development and preliminary psychometric testing of a new OA pain measure--an OARSI/OMERACT initiative. Osteoarthritis Cartilage. 2008 Apr;16(4):409-14. doi: 10.1016/j.joca.2007.12.015. PMID 18381179
- [Background] Perruccio AV, Stefan Lohmander L, Canizares M, Tennant A, Hawker GA, Conaghan PG, Roos EM, Jordan JM, Maillefert JF, Dougados M, Davis AM. The development of a short measure of physical function for knee OA KOOS-Physical Function Shortform (KOOS-PS) - an OARSI/OMERACT initiative. Osteoarthritis Cartilage. 2008 May;16(5):542-50. doi: 10.1016/j.joca.2007.12.014. Epub 2008 Feb 21. PMID 18294869